CLINICAL TRIAL: NCT02779179
Title: Efficacy of Therapeutic Management of Periodontitis on the Clinical Manifestations of Rheumatoid Arthritis: the Randomized, Controlled ESPERA Trial.
Brief Title: Therapeutic Management of Periodontitis and Clinical Manifestations of Rheumatoid Arthritis
Acronym: ESPERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10 046 08; 2010-A01193-36 (Registry Identifier: National Agency of Drug Safety and Health Products)
Record Dates: First submitted 2015-07-10; First posted 2016-05-20 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2018-11

CONDITIONS: Periodontitis; Rheumatoid Arthritis
MeSH Terms: conditions — Periodontitis; Arthritis, Rheumatoid | interventions — Periodontal Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Periodontal treatment group (Experimental)
  Interventions: Procedure: Periodontal treatment
- Delayed Periodontal treatment Group (Active Comparator)
  Interventions: Procedure: Periodontal treatment

INTERVENTIONS:
Procedure: Periodontal treatment — * Mechanical debridement (scaling, root planning, subgingival curettage)
  * Antimicrobial therapy (systematically administered: amoxicillin or clindamycin).
  * Antiseptic mouthrinses, gel or dentifrice
  * Oral hygiene instructions (to educate and motivate patients to control the accumulation of plaque and calculus)

SUMMARY:
Although RA pathomechanisms remains incompletely understood, periodontitis and RA share pathogenic features : genetic and environmental influences, chronic inflammatory disease, immunoregulatory imbalance, bacterial factors, persistence of antigen/peptide and clinical factors (conjunctive and hard tissues destruction). Several hypothesis can be evocated : Gram negative bacterial systemic spreading, inflammatory transmitter substance systemic spreading (IL1, IL6, IL17, PGE2), systemic spreading of bacterial degradation products (LPS for example).

Currently Porphyromonas gingivalis (PG) might be a susceptibility factor to RA because PG has an enzyme, the peptidylarginine deiminase leading to auto antibodies creation and RA increasing. As periodontitis, RA is chronic disease with a cyclic increase evolution, needing a complex pluridisciplinary treatment approach. Recent studies have reported an increased prevalence of RA patients with periodontal disease. Others studies show that periodontal treatment induces a significant decrease of the sedimentation rate and of the DAS28. Periodontitis is suspected to be an independent, aggravating factor in patients with RA (given the definition from NIH : an aggravating factor is something that makes a condition worse). So periodontal treatment cannot be considered as a RA treatment per se. But it is hypothesised that treating periodontitis in RA patients showing signs of periodontitis could result in improvement in RA disease activity. To date the role of periodontitis as an aggravating factor in these patients remains unclear, and only RCT designs can reasonably be used to test this causal hypothesis. There still remains some RA patients who have persistent symptoms and frequent exacerbations despite specialist care and continuous treatment, so results of treating aggravating factors are needed. As the majority of patients will benefit from a systematic evaluation and treatment of aggravating factors, the periodontal treatment strategy need to be tested.

The aim of this randomised controlled trial is to assess the effectiveness of periodontal treatment for rheumatoid arthritis patients.

To assess the effectiveness of periodontal treatment to reduce the severity of rheumatoid arthritis (RA), in patients suffering from both periodontitis and rheumatoid arthritis. The hypothesis is that periodontal treatment reduce the severity of rheumatoid arthritis.

ELIGIBILITY:
INCLUSION CRITERIA:

* rheumatoid arthritis diagnosed for at least one year
* DAS28 score between 3.2 and 5.1
* no change to medication, dosage or formulation in RA treatment during the 3 months preceding the screening visit
* subject available for all study visits over three months in the Dental Care Departments (V1 to V4)
* subjects with at least six natural teeth with root
* subject with periodontitis, defined by the presence of one site with periodontal probing depth ≥ 4 mm and clinical attachment level ≥ 3 mm on at least 4 teeth.
* subject has given his informed consent: 1 week cooling-off period

EXCLUSION CRITERIA:

* subject will not qualify for enrolment if he presents at least one of the following: acute oral infection, acute oral pain (including pulpitis), suspicious oral mucosal lesion, severe oral inflammation unrelated to periodontal conditions, or need for immediate tooth extractions
* have a planned hospitalization within 4 months after the screening visit
* subject suffering from one or more known infectious diseases (HIV, hepatitis, infectious mononucleosis),
* subject suffering from known clinically significant renal disease (creatinine clearance <60 ml/min), or liver disease,
* unbalanced diabetes
* have a known risk of endocarditis,
* have a permanent pacemaker,
* subject taking antithrombotic treatment,
* subject having severe difficulties in understanding written and spoken French
* for females: are pregnant or intending to become pregnant, or lactating
* subject suffering from a chronic disorder that requires chronic or intermittent use of antibiotics,
* subject having known hypersensitivity to chlorhexidine gluconate
* are participating in another intervention study
* have known contraindications to both amoxicillin and clindamycin
* have known contraindications to dental local anesthetic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of parodontitis therapeutic care as assessed by variation in DAS28 score | Day 15 and day 90

SECONDARY OUTCOMES:
Evaluation of parodontitis therapeutic care as assessed by variation in ACR 20 score | Day 15 and day 90
Evaluation of parodontitis therapeutic care as assessed by variation in HAQ score | Day 15 and day 90
Evaluation of parodontitis therapeutic care as assessed by variation in GOHAI score | Day 15 and day 90

CONTACTS AND LOCATIONS:
Overall Officials: Paul MONSARRAT, MD, Principal Investigator — Faculté de chirurgie dentaire - Toulouse
Locations (2):
- France (2):
  - CHU de Bordeaux, Bordeaux
  - Pôle Odontologie Hôpital Purpan - Pavillon Rayer, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Monsarrat P, Vergnes JN, Cantagrel A, Algans N, Cousty S, Kemoun P, Bertrand C, Arrive E, Bou C, Sedarat C, Schaeverbeke T, Nabet C, Sixou M. Effect of periodontal treatment on the clinical parameters of patients with rheumatoid arthritis: study protocol of the randomized, controlled ESPERA trial. Trials. 2013 Aug 14;14:253. doi: 10.1186/1745-6215-14-253. PMID 23945051
- [Result] Monsarrat P, Fernandez de Grado G, Constantin A, Willmann C, Nabet C, Sixou M, Cantagrel A, Barnetche T, Mehsen-Cetre N, Schaeverbeke T, Arrive E, Vergnes JN; ESPERA Group. The effect of periodontal treatment on patients with rheumatoid arthritis: The ESPERA randomised controlled trial. Joint Bone Spine. 2019 Oct;86(5):600-609. doi: 10.1016/j.jbspin.2019.02.006. Epub 2019 Feb 26. PMID 30822490